# Understanding Participation Habits: An Observational Investigation within Semantic Dementia Clinical Trials

An Informed Consent Form For Power Clinical Trial's
Observational Research on Semantic Dementia Clinical Trials
Patients

Date: January 12, 2024

Introduction to the Informed Consent Document: A Concise Overview

This summary is crafted to present a snapshot of our observational clinical study, focusing on its processes, potential risks, and benefits for participants. While your consent is mandatory, your involvement is entirely voluntary, allowing you the freedom to withdraw without any negative implications.

Our study seeks to fathom the reasons influencing individuals with semantic dementia in their decisions to enroll, persist, or discontinue participation in clinical trials. The primary procedures encompass the completion of questionnaires and follow-up calls, meticulously designed to minimize potential risks for participants.

Although immediate medical benefits may not be apparent in this observational study, the compiled data will play a pivotal role in pinpointing strategies to enhance clinical trial participation rates, ultimately benefiting those grappling with semantic dementia.

The study's findings will furnish vital insights into the determinants of clinical trial participation rates. Our goal is to refine recruitment strategies and reinforce patient engagement in trials, contributing to enhanced treatment options and outcomes for those with semantic dementia. Remember, participation is voluntary, and opting out will not impact your rights.

It is imperative to thoroughly scrutinize the consent form and seek clarification on any concerns before deciding. Engaging in discussions with family, friends, advisors, and healthcare professionals is recommended to ensure an informed choice. Participation remains voluntary. You can withdraw at any time without facing consequences.

Influential Factors in Semantic Dementia Clinical Trial Participation

Clinical trials are pivotal for advancing semantic dementia treatments, yet there are persistent concerns about participant diversity. This study seeks to unravel the determinants shaping patient decisions regarding participation, withdrawal, or re-engagement in semantic dementia clinical trials. Uncovering these factors is essential to enhance the relevance and efficacy of future research initiatives.

Our approach emphasizes a comprehensive understanding by recruiting a diverse demographic pool. We aim to decipher how variables such as age, race, income, and education influence decisions about participation. The collected data aims to craft more effective approaches to engage underrepresented groups in upcoming clinical trials.

Participation in this study is entirely voluntary, providing individuals with the liberty to withdraw without consequences. The study's procedures, involving questionnaire completion and follow-up calls, present minimal risks. Prospective participants are strongly encouraged to thoroughly review the consent form and seek clarification for any queries.

In essence, this trial seeks to deepen our understanding of the factors influencing semantic dementia clinical trial participation. Boosting participation rates could expedite the development of innovative treatments for this challenging condition.

Exploring Participation Behavior of Individuals with Semantic in Clinical Trials

Our observational clinical research endeavors to understand the nuanced factors guiding individuals with semantic dementia in their decisions related to clinical trial participation—be it enrollment, withdrawal, or completion. To identify potential participants, we seek involvement from those in ongoing or concluded interventional trials, utilizing electronic medical records for identification.

Upon expressing interest, our team provides a comprehensive consent form elucidating the study's objectives and participant rights. The data collection process involves regular biweekly questionnaires that delve into demographics, medical history, and the motivations influencing trial participation. Additionally, we plan to conduct thorough quarterly phone or video interviews to gain profound insights from participants.

The statistical analysis of the amassed data seeks to unveil the diverse factors influencing patient participation in clinical trials. Disseminating our findings through conferences and academic publications is geared toward benefiting all stakeholders involved in clinical trials.

These insights aim to inform the design of future clinical studies for individuals with semantic dementia, refining recruitment strategies and ensuring improved retention rates.

Participation in this study is entirely voluntary, providing individuals the liberty to withdraw without facing any consequences. The minimal risks involve the completion of questionnaires and follow-up interviews, with our readily accessible research team available to promptly address any queries or concerns.

Exploring Potential Risks in Observational Studies on Semantic Dementia

Participating in observational studies centered around semantic dementia doesn't involve experimental treatments, yet it may present certain risks. These risks may encompass breaches of privacy, emotional distress arising from the study's subject matter, and potential negative consequences from trial-related procedures.

Before making a decision to participate, it is imperative to meticulously scrutinize and understand the informed consent form and address any concerns with the research team. The team is dedicated to furnishing comprehensive information regarding potential risks, the study's benefits, and the safety measures implemented to safeguard the well-being of participants.

Unveiling the Potential Advantages of Semantic Dementia Observational Trials

Engaging in observational clinical trials dedicated to semantic dementia provides patients with a platform to contribute to medical advancements and potentially shape future treatment alternatives. Even in the absence of experimental therapies, participants can benefit from comprehensive care throughout the study.

Before committing to trial participation, patients are advised to thoroughly weigh potential benefits and risks, factoring in their individual situations and aspirations. Seeking guidance from healthcare providers and the research team is pivotal for making a thoughtful and informed decision.

### Essential Factors Impacting the Decision to Conclude Your Participation

Acknowledging the possibility that your participation in a clinical trial might cease without explicit consent is a crucial consideration. Researchers or sponsors may decide to conclude the trial for various reasons, including study suspension, discontinuation of funding, or if it's deemed beneficial for your welfare.

Additionally, your participation could come to an end due to declining health, pregnancy, opting out following substantial updates, or failure to adhere to study guidelines. Reflecting on these factors thoughtfully before choosing to participate in a clinical trial is paramount.

# **Exploring Semantic Dementia Clinical Trials**

Participation in clinical trials for semantic dementia is entirely voluntary, granting participants the liberty to withdraw without facing adverse consequences.

For a comprehensive view of global <u>research on semantic dementia</u>, clinicaltrials.gov, overseen by the National Institutes of Health (NIH), stands as a vast repository of ongoing trials. Users have the flexibility to customize their search based on location and specific medical conditions.

Additionally, Power's reference page provides an up-to-date compilation of currently active <u>semantic dementia clinical trials</u> actively seeking participants.

## Exploring Online Avenues for Clinical Trial Diversity

Various online platforms cater to individuals seeking in-depth insights into clinical trial diversity. Here are a couple of articles that might pique your interest:

Taran, F. Andrei, Haywood L. Brown, and Elizabeth A. Stewart. "Racial diversity in uterine leiomyoma clinical studies." *Fertility and sterility* 94, no. 4 (2010): 1500-1503.

Clark, Luther T., Laurence Watkins, Ileana L. Piña, Mary Elmer, Ola Akinboboye, Millicent Gorham, Brenda Jamerson et al. "Increasing diversity in clinical trials: overcoming critical barriers." *Current problems in cardiology* 44, no. 5 (2019): 148-172.

These resources offer valuable insights into the challenges associated with clinical trial diversity and potential strategies to enhance inclusivity within research studies.

## Keeping Research Studies Confidential

Our primary goal is to keep the data obtained for this study secret. Although perfect secrecy cannot be guaranteed, strong safeguards have been put in place to protect it. Please keep in mind that legal duties may require the sharing of personal information. However, any study papers or presentations will emphasize your anonymity by not revealing your name or any personally identifying information.

Accrediting bodies, government regulatory agencies (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives may have access to your medical information for research, quality assurance, and data analysis reasons.

In unusual circumstances, we may require an "Authorization Form" explaining the use and sharing of your information for this project. Explicit authorization will be obtained before sharing your information or research samples with Power researchers, other academic institutions, or external commercial firms for future study. Your private information will be treated securely and safely destroyed when needed.

# Consent Agreement Recognition: Embracing the Terms

By affixing your signature to this consent agreement, you acknowledge and embrace the following stipulations:

- Comprehensive reading and understanding of this informed consent form, with encouragement to explore alternative perspectives before reaching a decision.
- Resolution of all your queries concerning the research project and its methodologies, ensuring you possess the requisite information for study participation.
- Thoughtful consideration of potential benefits, drawbacks, and alternatives associated with your participation in the research.
- Assurance that your voluntary engagement in the research study will not encumber your legal rights.
- Timely communication of any substantial updates that may influence your decision to continue participating in the research study.
- Receipt of this consent form empowers you to address any lingering inquiries.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Researcher's Affirmation | | |
| n my capacity as the researcher, I<br>promoting a thorough understanding<br>patient's participation is voluntary a | ng of the study. Additionally, I ha | • |
| Signature of Researcher Who | Received Consent | |

Name of Investigator

Signature of Investigator Date